CLINICAL TRIAL: NCT01329042
Title: Efficacy of Potassium Sodium Hydrogen Citrate Therapy on Renal Stone Recurrence and/or Residual Fragments After Shockwave Lithotripsy and Percutaneous Nephrolithotomy in Calcium Oxalate Urolithiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ouiheng International Healthcare Co., Ltd (Industry)
Collaborators: Chiang Mai University (Other); Prince Songkla University (Unknown); Chulalongkorn University (Other); Siriraj Hospital (Other)
Responsible Party: Bannakij Lojanapiwat, Division of urology, Department of surgery, Chiangmai University, Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UU01/47
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Kidney Calculi
Keywords: Potassium sodium citrate; stone recurrence; ESWL; PCNL; Hypocitraturia; intervention
MeSH Terms: conditions — Kidney Calculi | interventions — magnesium citrate, potassium citrate, pyridoxine HCl, sodium citrate drug combination; Citrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Potassium-sodium citrate — The treated group was given oral potassium-sodium citrate 81 mEq/day The control group received no treatment
  Other Names: Uralyt-U

SUMMARY:
Extracorporeal shock wave lithotripsy (ESWL) and Percutaneous nephrolithotomy (PCNL) become the therapy of choice for renal stone. Although providing good results, stone recurrence is usually found as the therapies do not change the underlying metabolic abnormality. Among the metabolic disorders, hypocitraturia is an important risk factor for calcium nephrolithiasis. This study evaluate the preventive effects of potassium sodium citrate on stone recurrence as well as stone growth post ESWL or PCNL, in patients with calcium-containing stones.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* stone free or had residual calcium oxalate stone fragments with a less than 4 mm. diameter at eight weeks after ESWL or PCNL

Exclusion Criteria:

* renal tubular obstruction
* serum creatinine > 2 mg/dl
* urinary tract infection (bacteria > 100,000 in urine culture)
* hypersensitive or contraindication to Potassium sodium hydrogen citrate
* insertion Double-J Stent
* history of arrhythmia, myocardial infarction or digitalis administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-05; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
rate of stone recurrence or stone growth | 12 months
  The patients were evaluated at 6 months after the initial treatment for serum chemistry and urinalysis. After 12 months, all patients were evaluated for serum chemistry, urinalysis, 24-hour urine study and plain KUB.

CONTACTS AND LOCATIONS:
Overall Officials: Bannakij Lojanapiwat, MD, Principal Investigator — Division of Urology, Department of Surgery, Chiangmai University, Thailand